CLINICAL TRIAL: NCT02055547
Title: A Single and Multiple-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8521 in Subjects
Brief Title: A Single and Multiple-Dose Study of MK-8521 in Healthy and Obese Males (MK-8521-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8521-002; 2013-000083-28 (EudraCT Number); MK-8521-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parts 1 and 2 were parallel in design and Part 3 was crossover in design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (19):
- Part 1 - Panel A - MK-8521 100μg > PBO (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 100μg in the first treatment period, and matching placebo (PBO) in the second treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 100μg; Drug: Placebo
- Part 1 - Panel A - PBO > MK-8521 300μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of PBO in the first treatment period, and MK-8521 300μg in the second treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 300μg; Drug: Placebo
- Part 1 - Panel A - MK-8521 100μg > MK-8521 300μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 100μg in the first treatment period, and MK-8521 300μg in the second treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 100μg; Drug: MK-8521 300μg
- Part 1 - Panel B - MK-8521 150μg > PBO > MK-8521 175μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 150μg in the first treatment period, PBO in the second treatment period, and MK-8521 175μg in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 150μg; Drug: MK-8521 175μg; Drug: Placebo
- Part 1- Panel B- MK-8521 150μg > MK-8521 200μg > MK-8521 175μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 150μg in the first treatment period, MK-8521 200μg in the second treatment period, and MK-8521 175μg in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 150μg; Drug: MK-8521 175μg; Drug: MK-8521 200μg
- Part 1 - Panel B - MK-8521 150μg > MK-8521 200μg > PBO (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 150μg in the first treatment period, MK-8521 200μg in the second treatment period, and PBO in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 150μg; Drug: MK-8521 200μg; Drug: Placebo
- Part 1 - Panel B - PBO > MK-8521 200μg > MK-8521 175μg (Experimental): Healthy male participants of 18 to 45 years of age received PBO in the first treatment period, MK-8521 200μg in the second treatment period, and MK-8521 175μg in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 175μg; Drug: MK-8521 200μg; Drug: Placebo
- Part 2 - Panel C - MK-8521 50μg > MK-8521 72μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 50μg Days 1 to 5 and MK-8521 72μg Days 6 to 10 in a single treatment period.
  Interventions: Drug: MK-8521 50/72μg
- Part 2 - Panel D - MK-8521 100μg > MK-8521 150μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 100μg Days 1 to 5 and MK-8521 150μg Days 6 to 10 in a single treatment period.
  Interventions: Drug: MK-8521 100μg; Drug: MK-8521 100/150μg
- Part 2 - Panel E - MK-8521 125μg > MK-8521 150μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 125μg Days 1 to 5 and MK-8521 150μg Days 6 to 10 in a single treatment period.
  Interventions: Drug: MK-8521 125μg; Drug: MK-8521 125/150μg
- Part 2 - Panel F - MK-8521 72μg > MK-8521 125μg (Experimental): Obese male participants of 45 to 65 years of age received a single dose of MK-8521 72μg Days 1 to 7 and MK-8521 125μg Days 8 to 14 in a single treatment period.
  Interventions: Drug: MK-8521 125μg; Drug: MK-8521 72/125μg
- Part 2 - Panels C+D+E - Pooled Placebo (Placebo Comparator): Healthy male participants of 18 to 45 years of age received PBO once daily for 10 days.
  Interventions: Drug: Placebo
- Part 2 - Panel F - Placebo (Placebo Comparator): Obese male participants of 45 to 65 years of age received a single dose of PBO Days 1 to 14.
  Interventions: Drug: Placebo
- Part 3 - Panel H - MK-8521 125μg > MK-8521 35μg > PBO (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 125μg (high dose) in the first treatment period, MK-8521 35μg (low dose) in the second treatment period, and PBO in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo
- Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 35μg (low dose) in the first treatment period, PBO MK-8521 in the second treatment period, and 125μg (high dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo
- Part 3 - Panel H - PBO > MK- 8521 125μg > MK-8521 35μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of PBO in the first treatment period, MK- 8521 125μg (high dose) in the second treatment period, and MK-8521 35μg (low dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo
- Part 3 - Panel H - PBO > MK- 8521 35μg > MK-8521 125μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of PBO in the first treatment period, MK- 8521 35μg (low dose) in the second treatment period, and MK-8521 125μg (high dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo
- Part 3 - Panel H - MK-8521 125μg > PBO > MK-8521 35μg (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 125μg (high dose) in the first treatment period, PBO in the second treatment period, and MK-8521 35μg (low dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo
- Part 3 - Panel H - MK-8521 35μg > MK-8521 125μg > PBO (Experimental): Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 35μg (low dose) in the first treatment period, MK-8521 125μg (high dose) in the second treatment period, and PBO in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
  Interventions: Drug: MK-8521 35μg; Drug: MK-8521 125μg; Drug: Placebo

INTERVENTIONS:
Drug: MK-8521 35μg — Single dose 35μg subcutaneous (SC) injection in a treatment period (Part 3, Panel H)
  Arms: Part 3 - Panel H - MK-8521 125μg > MK-8521 35μg > PBO; Part 3 - Panel H - MK-8521 125μg > PBO > MK-8521 35μg; Part 3 - Panel H - MK-8521 35μg > MK-8521 125μg > PBO; Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg; Part 3 - Panel H - PBO > MK- 8521 125μg > MK-8521 35μg; Part 3 - Panel H - PBO > MK- 8521 35μg > MK-8521 125μg
Drug: MK-8521 100μg — Single dose 100μg SC injection in a treatment period (Part 1, Panel A) and (Part 2, Panel D)
  Arms: Part 1 - Panel A - MK-8521 100μg > MK-8521 300μg; Part 1 - Panel A - MK-8521 100μg > PBO; Part 2 - Panel D - MK-8521 100μg > MK-8521 150μg
Drug: MK-8521 125μg — Single dose 125μg SC injection in a treatment period (Part 2, Panel E) and (Part 3, Panel H)
  Arms: Part 2 - Panel E - MK-8521 125μg > MK-8521 150μg; Part 2 - Panel F - MK-8521 72μg > MK-8521 125μg; Part 3 - Panel H - MK-8521 125μg > MK-8521 35μg > PBO; Part 3 - Panel H - MK-8521 125μg > PBO > MK-8521 35μg; Part 3 - Panel H - MK-8521 35μg > MK-8521 125μg > PBO; Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg; Part 3 - Panel H - PBO > MK- 8521 125μg > MK-8521 35μg; Part 3 - Panel H - PBO > MK- 8521 35μg > MK-8521 125μg
Drug: MK-8521 150μg — Single dose 150μg SC injection in a treatment period (Part 1, Panel B)
  Arms: Part 1 - Panel B - MK-8521 150μg > MK-8521 200μg > PBO; Part 1 - Panel B - MK-8521 150μg > PBO > MK-8521 175μg; Part 1- Panel B- MK-8521 150μg > MK-8521 200μg > MK-8521 175μg
Drug: MK-8521 175μg — Single dose 175μg SC injection in a treatment period (Part 1, Panel B)
  Arms: Part 1 - Panel B - MK-8521 150μg > PBO > MK-8521 175μg; Part 1 - Panel B - PBO > MK-8521 200μg > MK-8521 175μg; Part 1- Panel B- MK-8521 150μg > MK-8521 200μg > MK-8521 175μg
Drug: MK-8521 200μg — Single dose MK-8521 200μg SC injection in a treatment period (Part 1, Panel B)
  Arms: Part 1 - Panel B - MK-8521 150μg > MK-8521 200μg > PBO; Part 1 - Panel B - PBO > MK-8521 200μg > MK-8521 175μg; Part 1- Panel B- MK-8521 150μg > MK-8521 200μg > MK-8521 175μg
Drug: MK-8521 300μg — Single dose 300μg SC injection in a treatment period (Part 1, Panel A)
  Arms: Part 1 - Panel A - MK-8521 100μg > MK-8521 300μg; Part 1 - Panel A - PBO > MK-8521 300μg
Drug: MK-8521 50/72μg — MK-8521 50μg SC injection Days 1-5 and 72μg Days 6-10 (Part 2, Panel C)
  Arms: Part 2 - Panel C - MK-8521 50μg > MK-8521 72μg
Drug: MK-8521 72/125μg — MK-8521 72μg SC injection Days 1-7 and 125μg Days 8-14 (Part 2, Panel F)
  Arms: Part 2 - Panel F - MK-8521 72μg > MK-8521 125μg
Drug: MK-8521 100/150μg — MK-8521 100μg SC injection Days 1-5 and 150μg Days 6-10 SC in a treatment period (Part 2, Panel D)
  Arms: Part 2 - Panel D - MK-8521 100μg > MK-8521 150μg
Drug: MK-8521 125/150μg — MK-8521 SC 125μg SC injection Days 1-5 and 150μg Days 6-10 (Part 2, Panel E)
  Arms: Part 2 - Panel E - MK-8521 125μg > MK-8521 150μg
Drug: Placebo — Placebo to MK-8521 SC injection in a treatment period (Parts 1, 2, and 3)
  Arms: Part 1 - Panel A - MK-8521 100μg > PBO; Part 1 - Panel A - PBO > MK-8521 300μg; Part 1 - Panel B - MK-8521 150μg > MK-8521 200μg > PBO; Part 1 - Panel B - MK-8521 150μg > PBO > MK-8521 175μg; Part 1 - Panel B - PBO > MK-8521 200μg > MK-8521 175μg; Part 2 - Panel F - Placebo; Part 2 - Panels C+D+E - Pooled Placebo; Part 3 - Panel H - MK-8521 125μg > MK-8521 35μg > PBO; Part 3 - Panel H - MK-8521 125μg > PBO > MK-8521 35μg; Part 3 - Panel H - MK-8521 35μg > MK-8521 125μg > PBO; Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg; Part 3 - Panel H - PBO > MK- 8521 125μg > MK-8521 35μg; Part 3 - Panel H - PBO > MK- 8521 35μg > MK-8521 125μg

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of MK-8521.

Part 1 primary hypothesis: Administration of single subcutaneous (SC) doses of MK-8521 is sufficiently safe and well- tolerated in healthy participants, based on assessment of clinical and laboratory adverse experiences, to permit continued clinical investigation.

Part 2: Administration of multiple once daily SC doses of MK-8521 is sufficiently safe and well-tolerated in healthy lean and obese participants, based on assessment of clinical and laboratory adverse experiences, to permit continued clinical investigation.

DETAILED DESCRIPTION:
This was a 3 part, randomized, single and multiple ascending-dose trial that evaluated the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of MK-8521 in healthy non-obese male (Part 1-Panels A and B, Panels C, D, and E of Part 2, and Part 3 Panel H) participants between the ages of 18 and 45 years and obese male participants (Part 2, Panel F) 45 to 65 years of age. An optional Panel G in Part 2 per protocol did not occur.

Part 1 was a single rising dose study to assess the safety and pharmacokinetics of single subcutaneous (SC) doses of MK-8521. Two panels of 8 healthy young non-obese male participants were dosed in up to 3 alternating dosing periods of MK-8521 or placebo (in a 6:2 ratio). Participants had a minimum 7 day washout between dosing periods.

Part 2 was a multiple-rising dose study to assess the safety and pharmacokinetics of multiple SC doses of MK-8521. Three panels (C-E) of 8 healthy young non-obese male participants received daily SC doses of MK-8521 or placebo (in a 6:2 ratio) as a titration regimen for 10 consecutive days. One panel (Panel F) of 8 older obese male participants received daily SC doses of MK-8521 or placebo (in a 6:2 ratio) as a titration regimen for 14 consecutive days.

Part 3 was a single dose, 3-period crossover study in 12 healthy lean male participants. Participants were randomized into 6 treatment groups and received a sequence of 3 treatments (MK-8521 at 35μg, 125μg and placebo). All participants in Part 3 received MK-8521 (high dose of 125μg and low dose of 35 μg) and placebo. There was a minimum 7 day washout between each dosing period for each individual participant.

ELIGIBILITY:
Inclusion Criteria:

* Males of either 18 to 45 or 45 to 70 years of age depending on the component of the study
* Body Mass Index between either 18-25 or 30-40 kg/m^2 depending on the component of the study
* Is in good health
* Is a non-smoker and/or has not used nicotine for at least 3 months

Exclusion Criteria:

* Is mentally or legally incapacitated, has significant emotional problems or has a history of psychiatric disorders in the past 5 years
* Has a history of the following abnormalities or diseases: endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological.
* History of cancer
* History of significant multiple or severe allergies or has had an anaphylactic reaction or significant intolerability to drugs or food
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Had major surgery, donated or lost 1 unit (500 mL) of blood or participated in another study within prior 4 weeks
* Has irritable bowel disease or recurrent nausea, vomiting, diarrhea or abdominal pain
* History of acute or chronic pancreatitis
* Uses 2 weeks prior to trial, or anticipates using during trial, medications, drugs or herbal remedies such as St. John's Wort
* Consumes greater than 3 glasses of alcohol per day
* Consumes greater than 6 servings of caffeinated beverages per day
* Regularly uses illicit drugs or has a history of drug (including alcohol) abuse within prior 3 months
* Has known hypersensitivity to glucagon or any glucagon like peptide 1 (GLP-1) receptor agonist
* Is unwilling/unable to consume standardized meals and/or is on a carbohydrate restricted diet
* Has history of hypersensitivity to pharmacologic insulins

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2013-09-17 (Actual); Study Completion 2013-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one clinical site in Belgium.
Pre-assignment Details: An optional Panel G in Part 2 per protocol did not occur.
  Period-level data were not collected for each treatment sequence.
Groups:
- Part 1 - Panel B - MK-8521 150μg > 200μg > MK-8521 175μg: Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 150μg in the first treatment period, MK-8521 200μg in the second treatment period, and MK-8521 175μg in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
- Part 2 - Panels C, D, and E - Pooled PBO: Healthy young lean male participants received matching placebo for MK-8521 once daily for 10 days.
- Part 2 - Panel F - MK-8521 72μg > MK-8521 125μg or PBO: Obese male participants of 45 to 65 years of age received a single dose of MK-8521 72μg Days 1 to 7 and MK-8521 125μg Days 8 to 14 or placebo in a single treatment period.
- Part 2 - Panel F - Placebo: Obese male participants of 45 to 65 years of age received a single dose of matching placebo for MK-8521 Days 1 to 14.
- Part 3 - Panel H - MK-8521 125μg > 35μg > PBO: Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 125μg (high dose) in the first treatment period, MK-8521 35μg (low dose) in the second treatment period, and PBO in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
- Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg: Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 35μg (low dose) in the first treatment period, PBO in the second treatment period, and 125μg (high dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
- Part 3 - Panel H - PBO > MK-8521 125μg > 35μg: Healthy male participants of 18 to 45 years of age received a single dose of PBO in the first treatment period, MK-8521 125μg (high dose) in the second treatment period, and MK-8521 35μg (low dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
- Part 3 - Panel H - PBO > MK-8521 35μg > 125μg: Healthy male participants of 18 to 45 years of age received a single dose of PBO in the first treatment period, MK-8521 35μg (low dose) in the second treatment period, and MK-8521 125μg (high dose) in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
- Part 3 - Panel H - MK-8521 35μg > 125μg > PBO: Healthy male participants of 18 to 45 years of age received a single dose of MK-8521 35μg (low dose) in the first treatment period, MK-8521 125μg (high dose) in the second treatment period, and PBO in the third treatment period. There was a minimum of a 7-day washout period between treatment periods.
Period: Overall Study
Arm/Group | Part 1 - Panel A - MK-8521 100μg > PBO | Part 1 - Panel A - PBO > MK-8521 300μg | Part 1 - Panel A - MK-8521 100μg > MK-8521 300μg | Part 1 - Panel B - MK-8521 150μg > PBO > MK-8521 175μg | Part 1 - Panel B - MK-8521 150μg > 200μg > MK-8521 175μg | Part 1 - Panel B - MK-8521 150μg > MK-8521 200μg > PBO | Part 1 - Panel B - PBO > MK-8521 200μg > MK-8521 175μg | Part 2 - Panel C - MK-8521 50μg > MK-8521 72μg | Part 2 - Panel D - MK-8521 100μg > MK-8521 150μg | Part 2 - Panel E - MK-8521 125μg > MK-8521 150μg | Part 2 - Panels C, D, and E - Pooled PBO | Part 2 - Panel F - MK-8521 72μg > MK-8521 125μg or PBO | Part 2 - Panel F - Placebo | Part 3 - Panel H - MK-8521 125μg > 35μg > PBO | Part 3 - Panel H - MK-8521 35μg > PBO > MK-8521 125μg | Part 3 - Panel H - PBO > MK-8521 125μg > 35μg | Part 3 - Panel H - PBO > MK-8521 35μg > 125μg | Part 3 - Panel H - MK-8521 125μg > PBO > MK-8521 35μg | Part 3 - Panel H - MK-8521 35μg > 125μg > PBO
Started | 2 | 2 | 5 | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 6 | 6 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 6 | 4 | 5 | 5 | 6 | 2 | 1 | 2 | 1 | 2 | 2 | 2
Not Completed | 0 | 1 | 3 | 0 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population included all treated study participants. Baseline characteristics were not captured in the study by individual treatment sequences.
Groups:
- Part 1 - 3, Panel A, B, C, D, E, F, and H: All participants who received a dose of MK-8521 or placebo in any study period.
Arm/Group | Part 1 - 3, Panel A, B, C, D, E, F, and H
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE) (Part 1)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: From Day 1 through post-trial visit (Up to 8 weeks)
Population: The analysis population included all participants in Part 1 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Panel A MK-8521 100μg: MK-8521 100μg in healthy male participants of 18 to 45 years of age
- Part 1 Panel A MK-8521 300μg: MK-8521 300μg in healthy male participants of 18 to 45 years of age
- Part 1 Panel B MK-8521 150μg: MK-8521 150μg in healthy male participants of 18 to 45 years of age
- Part 1 Panel B MK-8521 175μg: MK-8521 175μg in healthy male participants of 18 to 45 years of age
- Part 1 Panel B MK-8521 200μg: MK-8521 200μg in healthy male participants of 18 to 45 years of age
- Part 1, Pooled Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg | Part 1, Pooled Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5 | 16
Participants | 3 | 4 | 2 | 0 | 5 | 10

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE (Part 1)
Description: as for outcome 1
Time Frame: Up to 8 weeks (Part 1)
Population: The analysis population included all participants in Part 1 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg | Part 1, Pooled Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Area Under the Concentration Time Curve of MK-8521 From 0 to Infinity (AUC0-∞) After a Single Dose (Part 1)
Description: AUC0-∞ is a measure of the mean concentration levels of drug in the plasma after the dose. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part I, Panels A-B, Period 1-3 [100-300μg]) is presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24, 30, 34, 48, 72, 96, 120 hrs. post-dose (Part 1)
Population: The analysis population included a subset of participants in Part 1 who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hr
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5
nM•hr | 48.7 (16.4) | 163 (6.37) | 84.4 (20.3) | 101 (6.07) | 109 (25.7)

4. Primary Outcome: Peak Plasma Concentration (Cmax) of Participants Treated With a Single Dose of MK-8521 (Part 1)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part I, Panels A-B, Period 1-3 [100-300μg]) is presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24, 30, 34, 48, 72, 96, 120 hrs. post-dose (Part 1)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5
nM | 1.24 (30.2) | 4.29 (23.5) | 2.63 (20.0) | 3.10 (20.8) | 3.54 (18.4)

5. Primary Outcome: Time Taken to Reach Cmax (Tmax) for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 1)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part I, Panels A-B, Period 1-3 [100-300μg]) is presented. No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24, 30, 34, 48, 72, 96, 120 hrs. post-dose (Part 1)
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5
Hours | 14 [8 to 30] | 10 [4 to 16] | 11 [10 to 16] | 12 [8 to 12] | 14 [10 to 16]

6. Primary Outcome: Apparent Terminal Half-life (t1/2) for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 1)
Description: Apparent Terminal Half-life (t1/2) is the time required for a given drug concentration in the plasma to decrease by 50%. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part I, Panels A-B, Period 1-3 [100-300μg]) is presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24, 30, 34, 48, 72, 96, 120 hrs. post-dose (Part 1)
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5
Hours | 13.8 (15.5) | 13.7 (8.93) | 14.8 (6.45) | 14.1 (2.64) | 13.8 (12.9)

7. Primary Outcome: Number of Participants With an Adverse Event (AE) (Part 2)
Description: as for outcome 1
Time Frame: From Day 1 through post-trial visit (Up to 7 weeks)
Population: The analysis population included all participants in Part 2 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2 Panel C MK-8521 50/72μg: MK-8521 50μg Days 1-5 and 72μg Days 6-10 or Placebo in healthy male participants of 18 to 45 years of age
- Part 2 Panel D MK-8521 100/150μg: MK-8521 100μg Days 1-5 and 150μg Days 6-10 in healthy male participants of 18 to 45 years of age
- Part 2 Panel E MK-8521 125/150μg: MK-8521 125μg Days 1-5 and 150μg Days 6-10 in healthy male participants of 18 to 45 years of age
- Part 2 Panel F MK-8521 72/125μg: MK-8521 72μg Days 1-7 and 125μg Days 8-14 in obese male participants of 45 to 65 years of age
- Part 2, Pooled Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg | Part 2 Panel F MK-8521 72/125μg | Part 2, Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 5 | 5 | 5 | 4 | 3

8. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE (Part 2)
Description: as for outcome 1
Time Frame: Up to 7 weeks (Part 2)
Population: The analysis population included all participants in Part 2 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg | Part 2 Panel F MK-8521 72/125μg | Part 2, Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 0 | 1 | 0 | 0 | 0

9. Primary Outcome: AUC 0-24hr for Plasma Concentration of Participants Treated After Multiple Doses of MK-8521 (Part 2, Panels C, D, and E)
Description: AUC0-24hr is a measure of the mean concentration levels of drug in the plasma 0 to 24 hrs. after the dose. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part II, Panel C, D, and E) are presented. Method of dispersion coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected at the following time points for Part 2, Panel C, D, and E: Days 1, 4, 5, 9, 10 pre-dose; Days 1, 5, 10: 2, 4, 8, 10, 12, 16, 24 hrs. post dose; Day 10: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 5 and 10 (Part 2) (Panels C, D, E)
Population: The analysis population included a subset of participants in Part 2 (Panels C, D, and E) who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hr
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg
Number analyzed (Participants) | 6 | 6 | 6
nM•hr
  Day 1 | 12.0 (21.3) | 23.1 (18.9) | 33.5 (16.4)
  Day 5 | 22.8 (20.7) | 43.3 (23.6) | 60.7 (19.8)
  Day 10: number analyzed (Participants) | 6 | 4 | 5
  Day 10 | 35.1 (19.0) | 86.8 (34.4) | 77.8 (15.0)

10. Primary Outcome: AUC 0-24hr for Plasma Concentration of Participants Treated After Multiple Doses of MK-8521 (Part 2, Panel F)
Description: AUC0-24hr is a measure of the mean concentration levels of drug in the plasma 0 to 24 hrs. after the dose. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 14 Days (with dose escalation on Day 7) to obese male participants (Part 2, Panel F) are presented. Method of dispersion coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected at the following time points for Part 2, Panel F: Days 1, 3, 4, 5, 7, 9, 11, 13, 14 pre-dose; Days 1, 7, 14: 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24 hrs. post-dose; Day 14: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 7 and 14 (Part 2) (Panel F)
Population: The analysis population included a subset of participants in Part 2 (Panel F) who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hr
Arm/Group | Part 2 Panel F MK-8521 72/125μg
Number analyzed (Participants) | 6
nM•hr
  Day 1 | 8.85 (22.1)
  Day 7 | 24.8 (21.6)
  Day 14 | 54.6 (17.9)

11. Primary Outcome: Cmax for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panels C, D, and E)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part 2, Panel C, D, E and F) are presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected at the following time points for Part 2, Panel C-E: Days 1, 4, 5, 9, 10 pre-dose; Days 1, 5, 10: 2, 4, 8, 10, 12, 16, 24 hrs. post dose; Day 10: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 5 and 10 (Part 2) (Panels C, D, E)
Population: The analysis population included participants in Part 2 (Panels C, D, and E) who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg
Number analyzed (Participants) | 6 | 6 | 6
nM
  Day 1 | 0.642 (21.8) | 1.25 (20.0) | 1.85 (23.1)
  Day 5 | 1.11 (22.6) | 2.21 (23.1) | 3.12 (16.0)
  Day 10: number analyzed (Participants) | 6 | 4 | 5
  Day 10 | 1.73 (20.4) | 4.31 (35.9) | 3.73 (13.0)

12. Primary Outcome: Cmax for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: as for outcome 10
Time Frame: Days 1, 7 and 14 (Part 2) (Panel F)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2 Panel F MK-8521 72/125μg
Number analyzed (Participants) | 6
nM
  Day 1 | 0.511 (22.7)
  Day 7 | 1.15 (22.8)
  Day 14 | 2.56 (19.6)

13. Primary Outcome: Trough Plasma Concentration (Ctrough) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panels C, D, and E)
Description: Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]). Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part 2, Panel C, D, and E) are presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected for Part 2, Panel C, D, and E: Days 1, 4, 5, 9, 10 pre-dose; Days 1, 5, 10: 2, 4, 8, 10, 12, 16, 24 hrs. post dose; Day 10: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 5 and 10 (Part 2) (Panels C, D, E)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg
Number analyzed (Participants) | 6 | 6 | 6
nM
  Day 1 | 0.493 (17.6) | 1.00 (25.0) | 1.33 (19.6)
  Day 5 | 0.721 (18.8) | 1.33 (30.0) | 2.01 (15.7)
  Day 10: number analyzed (Participants) | 6 | 4 | 5
  Day 10 | 1.20 (14.4) | 2.92 (40.5) | 2.82 (17.7)

14. Primary Outcome: Trough Plasma Concentration (Ctrough) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration]). Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 14 Days (with dose escalation on Day 7) to obese male participants (Part 2, Panel F) are presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected at the following time points for Part 2, Panel F: Days 1, 3, 4, 5, 7, 9, 11, 13, 14 pre-dose; Days 1, 7, 14: 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24 hrs. post-dose; Day 14: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 7 and 14 (Part 2) (Panel F)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2 Panel F MK-8521 72/125μg
Number analyzed (Participants) | 6
nM
  Day 1 | 0.498 (22.8)
  Day 7 | 0.935 (18.6)
  Day 14 | 2.09 (15.3)

15. Primary Outcome: Tmax for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panels C, D, and E)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part 2, Panel C, D, and E) are presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections for the determination of plasma MK-8521 concentrations were collected at the following time points for Part 2, Panel C, D, and E: Days 1, 4, 5, 9, 10 pre-dose; Days 1, 5, 10: 2, 4, 8, 10, 12, 16, 24 hrs. post dose; Day 10: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 5 and 10 (Part 2) (Panels C, D, E)
Population: The analysis population included participants in Part 2 (Panels C, D, and E) who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg
Number analyzed (Participants) | 6 | 6 | 6
Hours
  Day 1 | 12 [10 to 12] | 10 [8 to 24] | 10 [8 to 16]
  Day 5 | 9 [8 to 12] | 8 [8 to 12] | 9 [4 to 12]
  Day 10: number analyzed (Participants) | 6 | 4 | 5
  Day 10 | 8 [8 to 10] | 10 [10 to 12] | 10 [8 to 12]

16. Primary Outcome: Tmax for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 14 Days (with dose escalation on Day 7) to obese male participants (Part 2, Panel F) are presented. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 14 Days (with dose escalation on Day 7) to obese male participants (Part 2, Panel F) are presented. Method of dispersion is coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections occurred at the following time points for Part 2, Panel F: Days 1, 3, 4, 5, 7, 9, 11, 13, 14 pre-dose; Days 1, 7, 14: 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24 hrs. post-dose; Day 14: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 7 and 14 (Part 2) (Panel F)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2 Panel F MK-8521 72/125μg
Number analyzed (Participants) | 6
Hours
  Day 1 | 24 [12 to 24]
  Day 7 | 9 [8 to 10]
  Day 14 | 10 [8 to 16]

17. Primary Outcome: Apparent Terminal Half-life (t1/2) for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Part C, D, and E)
Description: Apparent Terminal Half-life (t1/2) is the time required for a given drug concentration in the plasma to decrease by 50%. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part 2, Panel C, D, and E) are presented. Method of dispersion is coefficient of variation (%CV). Apparent terminal t1/2 was not reported for certain days since the terminal phase was not adequately captured with sampling up to 24hr post dose. No pharmacokinetic analysis was performed on participants receiving Placebo. Blood was collected for Part 2, Panel C, D, and E: Days 1, 4, 5, 9, 10 pre-dose; Days 1, 5, 10: 2, 4, 8, 10, 12, 16, 24 hrs. post dose; Day 10: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 5 and 10 (Part 2) (Panels C, D, E)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg
Number analyzed (Participants) | 6 | 6 | 6
Hours
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 0 | 0 | 0
  Day 10 | 14.7 (17.7) | 15.9 (10.9) | 15.5 (12.5)

18. Primary Outcome: Apparent Terminal Half-life (t1/2) for Plasma Concentration of Participants Treated With Multiple Doses of MK-8521 (Part 2, Part F)
Description: Apparent Terminal Half-life (t1/2) is the time required for a given drug concentration in the plasma to decrease by 50%. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 14 Days (with dose escalation on Day 7) to obese male participants (Part 2, Panel F) are presented. Method of dispersion is coefficient of variation (%CV). Apparent terminal t1/2 was not reported for certain days since the terminal phase was not adequately captured with sampling up to 24hr post dose. No pharmacokinetic analysis was performed on participants receiving Placebo. Blood collections occurred at the following time points for Part 2, Panel F: Days 1, 3, 4, 5, 7, 9, 11, 13, 14 pre-dose; Days 1, 7, 14: 0.5, 1, 2, 4, 8, 10, 12, 14, 16, 24 hrs. post-dose; Day 14: 72, 96, 120 hrs. post-dose.
Time Frame: Days 1, 7 and 14 (Part 2) (Panel F)
Population: The analysis population included a subset of participants in Part 2 (Panels F) who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Groups:
- Part 2 Panel F MK-8521 72/125μgEdit: MK-8521 72μg Days 1-7 and 125μg Days 8-14 in obese male participants of 45 to 65 years of age
Arm/Group | Part 2 Panel F MK-8521 72/125μgEdit
Number analyzed (Participants) | 6
Hours
  Day 1: number analyzed (Participants) | 0
  Day 7: number analyzed (Participants) | 0
  Day 14 | 16.2 (8.4)

19. Primary Outcome: Number of Participants With an Adverse Event (AE) (Part 3)
Description: as for outcome 1
Time Frame: Up to 6 weeks (Part 3)
Population: The analysis population included all participants in Part 3 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 3 Panel H MK-8521 35μg: MK-8521 35μg in healthy male participants of 18 to 45 years of age
- Part 3 Panel H MK-8521 125μg: MK-8521 125μg in healthy male participants of 18 to 45 years of age
- Part 3, Pooled Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3, Pooled Placebo
Number analyzed (Participants) | 11 | 12 | 5
Participants | 5 | 8 | 3

20. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE (Part 3)
Description: as for outcome 1
Time Frame: Up to 6 weeks (Part 3)
Population: The analysis population included all participants in Part 3 who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3, Pooled Placebo
Number analyzed (Participants) | 11 | 12 | 5
Participants | 0 | 0 | 0

21. Primary Outcome: Average Concentration (Cave) of MK-8521 Corresponding to Slope of Insulin Secretion Rate/Glucose (ISR/G) During Graded Glucose Infusion (GGI) at Tmax After a Single Dose of MK-8521 (Part 3)
Description: Pancreatic beta cell sensitivity to ambient glucose concentration after a single dose of MK-8521 125μg/35μg or placebo at Tmax was quantified as the slope of insulin secretion rate relative to glucose concentration (ISR/G) during GGI (160 minutes duration) and assessed against MK-8521 average plasma concentration (Cave) during the GGI to preliminarily characterize the PK/ pharmacodynamic (PD) relationship. Study drug was administered on Day -1. Plasma concentrations of MK-8521 were determined at -10 min pre-GGI and 40, 80, 120 & 160 min and blood concentrations of glucose, insulin & C-peptide were determined at -10, -5 (pre-GGI), 20, 40, 60, 80, 100, 120, 140 & 160 minutes after start of GGI on Day 1 of each period. ISR calculated by deconvolution of C-peptide concentrations using a two-compartmental model was regressed on glucose concentration via simple linear regression; beta cell glucose sensitivity was defined as slope from the regression line.
Time Frame: From -10 to 160 minutes after GGI on Day 1 (Part 3)
Population: The analysis population included a subset of participants in Part 3 who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg
Number analyzed (Participants) | 11 | 12
nM | 0.376 (37.8) | 1.64 (24.4)

22. Secondary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hrs (TWA0-24hr) of Heart Rate (HR) After a Single Dose of MK-8521 (Part 1)
Description: Heart rate was assessed on Day 1 (predose & 1, 4, 8, 12, 16 & 24 hrs. postdose) & Day 2 (36 & 48 hrs. postdose). Predose and postdose HR were assessed using triplicate and duplicate measurements, respectively. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of HR on Day 1 & Day 2 of MK-8521 single dosing was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr HR was calculated for each participant where baseline was defined as predose baseline on Day 1.
Time Frame: Baseline (predose), up to 24 hours post-dose on Day 1, up to 24 hours post-dose on Day 2 (Part 1)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Groups:
- Part 1 - Pooled Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg | Part 1 - Pooled Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5 | 9
Beats per minute
  Day 1 | 6.67 [0.68 to 12.66] | 19.03 [12.30 to 25.76] | 0.06 [-6.32 to 6.44] | 9.28 [1.06 to 17.50] | 7.99 [1.17 to 14.81] | 2.76 [-2.43 to 7.95]
  Day 2 | 11.77 [5.78 to 17.76] | 20.91 [14.18 to 27.64] | 1.69 [-4.70 to 8.07] | 15.43 [7.22 to 23.65] | 13.73 [6.90 to 20.55] | 7.76 [2.56 to 12.95]

23. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Systolic Blood Pressure (SBP) of Participants Treated With A Single Dose of MK-8521 (Part 1)
Description: Systolic blood pressure was assessed on Day 1 (predose and 1, 4, 8, 12, 16 and 24 hrs. postdose) and Day 2 (36 and 48 hrs. postdose). Predose and postdose SBP were assessed using triplicate and duplicate measurements, respectively. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr. of SBP on Day 1 and Day 2 of MK-8521 single dosing was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr SBP was calculated for each participant where baseline was defined as predose baseline on Day 1.
Time Frame: Baseline (predose), up to 24 hours post-dose on Day 1, up to 24 hours post-dose on Day 2 (Part 1)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg | Part 1 - Pooled Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5 | 9
mmHg
  Day 1 | -1.09 [-5.67 to 3.50] | 8.43 [3.30 to 13.55] | -2.24 [-7.12 to 2.63] | 3.18 [-3.04 to 9.41] | 0.10 [-5.10 to 5.30] | 0.78 [-3.2 to 4.75]
  Day 2 | -2.55 [-7.14 to 2.03] | 7.81 [2.69 to 12.94] | -0.73 [-5.61 to 4.15] | 2.03 [-4.20 to 8.25] | 1.71 [-3.49 to 6.91] | 1.9 [-2.08 to 5.87]

24. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Diastolic Blood Pressure (DBP) of Participants Treated With A Single Dose of MK-8521 (Part 1)
Description: Diastolic blood pressure was assessed on Day 1 (predose and 1, 4, 8, 12, 16 & 24 hrs postdose) and Day 2 (36 and 48 hrs postdose). Predose and postdose DBP were assessed using triplicate and duplicate measurements, respectively. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of DBP on Day 1 and Day 2 of MK-8521 single dosing was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr DBP was calculated for each participant where baseline was defined as predose baseline on Day 1.
Time Frame: Baseline (predose), up to 24 hours post-dose on Day 1, up to 24 hours post-dose on Day 2 (Part 1)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part 1 Panel A MK-8521 100μg | Part 1 Panel A MK-8521 300μg | Part 1 Panel B MK-8521 150μg | Part 1 Panel B MK-8521 175μg | Part 1 Panel B MK-8521 200μg | Part 1 - Pooled Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 3 | 5 | 9
mmHg
  Day 1 | 0.30 [-3.85 to 4.46] | 5.60 [0.66 to 10.54] | -3.73 [-8.22 to 0.76] | -0.80 [-7.24 to 5.64] | 2.54 [-2.40 to 7.48] | -0.07 [-3.75 to 3.61]
  Day 2 | -1.41 [-5.56 to 2.75] | 5.55 [0.61 to 10.49] | -2.56 [-7.05 to 1.94] | 0.90 [-5.54 to 7.33] | 2.14 [-2.80 to 7.08] | 0.57 [-3.11 to 4.25]

25. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Heart Rate (HR) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel C, D, and E)
Description: Heart rate was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs post admission), Day 1 and Day 6 (predose and 2, 4, 6, 8, 12, 16, 24, 36 and 48 hrs postdose) and Day 10 (predose & 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose HR on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 6, and Day 10 HR were assessed using duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of HR on Day 1, Day 6, and Day 10 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs). The change from baseline TWA0-24hr HR was calculated for each participant using TWA0-24hr on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), predose & up to 24 hours postdose on Days 1, 6, and 10
Population: The analysis population included a subset of participants in Part 2, Panels C, D, and E who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Groups:
- Part 2 - Panel C, D, E - Pooled Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg | Part 2 - Panel C, D, E - Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Beats per minute
  Day 1 | 1.18 [-3.57 to 5.93] | 0.30 [-4.45 to 5.05] | 4.15 [-0.60 to 8.90] | -1.91 [-6.66 to 2.84]
  Day 6 | 4.24 [-0.51 to 8.99] | 7.96 [3.21 to 12.71] | 8.52 [3.77 to 13.27] | -0.74 [-5.49 to 4.01]
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | 9.30 [4.55 to 14.05] | 12.42 [7.67 to 17.17] | 9.88 [5.00 to 14.77] | 0.81 [-4.08 to 5.69]

26. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Heart Rate (HR) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: Heart rate was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs post admission), Day 1 & Day 8 (predose and 2, 4, 6, 8, 12, 16, 24, 36, and 48 hrs. post dose) & Day 14 (predose and 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose HR on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 8, and Day 14 HR were assessed as duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of HR on Day 1, Day 8, and Day 14 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr. HR was calculated for each participant using TWA0-24hr. on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), predose & up to 24 hours postdose on Days 1, 8, and 14
Population: The analysis population included a subset of participants in Part 2, Panel F who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment, according to the underlying scientific model. Compliance included exposure to treatment, availability of measurements, and absence of major protocol violations.
Measure: Mean (Standard Error); unit: Beats per minute
Groups:
- Part 2 - Panel F - Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 2 Panel F MK-8521 72/125μg | Part 2 - Panel F - Placebo
Number analyzed (Participants) | 6 | 2
Beats per minute
  Day 1 | 0.14 (1.33) | 0.52 (1.42)
  Day 8 | 5.22 (1.43) | 0.29 (0.66)
  Day 14 | 9.25 (2.14) | -1.11 (1.04)

27. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Systolic Blood Pressure (SBP) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panels C, D, and E)
Description: Systolic blood pressure was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs. post admission), Day 1 and Day 6 (predose & 2, 4, 6, 8, 12, 16, 24, 36, and 48 hrs. postdose) and Day 10 (predose & 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose SBP on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 6, and Day 10 SBP were assessed using duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr SBP on Day 1, Day 6 and Day 10 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs). The change from baseline TWA0-24hr SBP was calculated for each participant using TWA0-24hr on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), predose & up to 24 hours postdose on Days 1, 6, and 10
Population: as for outcome 25
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg | Part 2 - Panel C, D, E - Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmHg
  Day 1 | -0.12 [-3.87 to 3.63] | 1.57 [-2.18 to 5.31] | -2.65 [-6.40 to 1.09] | 1.19 [-2.56 to 4.93]
  Day 6 | -2.08 [-5.82 to 1.67] | -2.26 [-6.00 to 1.49] | -6.73 [-10.47 to -2.98] | -1.18 [-4.93 to 2.56]
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | -0.01 [-3.76 to 3.73] | -5.78 [-9.53 to -2.03] | -2.35 [-6.30 to 1.60] | -3.25 [-7.20 to 0.70]

28. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Systolic Blood Pressure (SBP) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: Systolic blood pressure was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs. post admission), Day 1 and Day 8 (predose and 2, 4, 6, 8, 12, 16, 24, 36, and 48 hrs. post dose) and Day 14 (predose and 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose SBP on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 8, and Day 14 SBP were assessed as duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of SBP on Day 1, Day 8, and Day 14 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr SBP was calculated for each participant using TWA0-24hr on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), up to 16 hrs on Day -1, predose & up to 24 hours postdose on Days 1, 8, and 14
Population: as for outcome 26
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Part 2 Panel F MK-8521 72/125μg | Part 2 - Panel F - Placebo
Number analyzed (Participants) | 6 | 2
mmHg
  Day 1 | -2.19 (2.33) | 1.82 (1.00)
  Day 8 | -3.99 (2.86) | -6.55 (0.24)
  Day 14 | -2.25 (4.15) | -9.43 (0.39)

29. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Diastolic Blood Pressure (DBP) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Part C, D, and E)
Description: Diastolic blood pressure was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs. post admission), Day 1 and Day 6 (predose and 2, 4, 6, 8, 12, 16, 24, 36 and 48 hrs. postdose) and Day 10 (predose and 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose DBP on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 6, and Day 10 DBP were assessed using duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr. DBP on Day 1, Day 6, and Day 10 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs.). The change from baseline TWA0-24hr DBP was calculated for each participant using TWA0-24hr. on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), predose & up to 24 hours postdose on Days 1, 6, and 10
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Part 2 Panel C MK-8521 50/72μg | Part 2 Panel D MK-8521 100/150μg | Part 2 Panel E MK-8521 125/150μg | Part 2 - Panel C, D, E - Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmHg
  Day 1 | 1.22 [-1.87 to 4.30] | 2.38 [-0.71 to 5.46] | 0.06 [-3.02 to 3.15] | 0.25 [-2.83 to 3.33]
  Day 6 | 0.37 [-2.71 to 3.46] | 2.63 [-0.45 to 5.72] | -1.22 [-4.31 to 1.86] | 0.68 [-2.41 to 3.76]
  Day 10: number analyzed (Participants) | 6 | 6 | 5 | 5
  Day 10 | 1.58 [-1.50 to 4.67] | 0.56 [-2.52 to 3.65] | 3.29 [0.09 to 6.50] | 0.53 [-2.67 to 3.74]

30. Secondary Outcome: Change From Baseline in TWA 0-24 Hrs. Semi-recumbent Diastolic Blood Pressure (DBP) of Participants Treated With Multiple Doses of MK-8521 (Part 2, Panel F)
Description: Diastolic blood pressure was assessed on Day -1 (at 2, 4, 6, 8, 12, and 16 hrs. post admission), Day 1 and Day 8 (predose and 2, 4, 6, 8, 12, 16, 24, 36, and 48 hrs. post dose) and Day 14 (predose and 2, 4, 6, 8, 12, 16, and 24 hrs. postdose). Predose DBP on Day 1 was assessed using triplicate measurements while Day -1, Day 1 (postdose), Day 8, and Day 14 DBP were assessed as duplicate measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr of DBP on Day 1, Day 8, Day 14 of MK-8521 multiple dose treatment was calculated as the area under the measurement-time curve divided by the time period of over which the measurements were made (i.e., 24 hrs). The change from baseline TWA0-24hr. DBP was calculated for each participant using TWA0-24hr. on Day -1 as the baseline.
Time Frame: Baseline (predose; up to 16 hrs on Day -1), predose & up to 24 hours postdose on Days 1, 8, and 14
Population: as for outcome 26
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Part 2 Panel F MK-8521 72/125μg | Part 2 - Panel F - Placebo
Number analyzed (Participants) | 6 | 2
mmHg
  Day 1 | -0.15 (1.30) | 1.45 (1.43)
  Day 8 | 0.41 (1.54) | -2.63 (1.11)
  Day 14 | 0.78 (2.32) | -3.19 (0.30)

31. Secondary Outcome: Slope of Insulin Secretion Rate/Glucose (ISR/G) During Graded Glucose Infusion (GGI) at Tmax After a Single Dose of MK-8521 (Part 3)
Description: Pancreatic beta cell sensitivity to ambient glucose concentration after a single dose of MK-8521 125μg/35μg or placebo at Tmax was quantified as the slope of insulin secretion rate relative to glucose concentration (ISR/G) during GGI (160 minutes duration). Study drug was administered on Day -1 and blood concentrations of glucose, insulin & C-peptide were determined at -10, -5 (pre-GGI), 20, 40, 60, 80, 100, 120, 140, and 160 minutes after start of GGI on Day 1 of each period. ISR calculated by deconvolution of C-peptide concentrations using a two compartmental model was regressed on glucose concentration via simple linear regression; beta cell glucose sensitivity was defined as slope from the regression line.
Time Frame: From -10 to 160 minutes after GGI on Day 1
Population: as for outcome 26
Measure: Least Squares Mean (95% Confidence Interval); unit: (ng/min.)/(mg/dL)
Groups:
- Part 3 - Panel H - Placebo: Healthy male participants of 18 to 45 years of age received PBO.
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 11
(ng/min.)/(mg/dL) | 0.0314 [0.024 to 0.0412] | 0.0543 [0.0417 to 0.0706] | 0.0118 [0.009 to 0.0154]
Statistical Analysis 1: Comparison: Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — Treatment comparison (MK-8521 125μg - placebo) of the slope of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of the slope of ISR/G for MK-8521 125μg vs. placebo was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 4.61, 90% CI 2-sided [3.69 to 5.76]; Number of participants included in analysis: N=17 (3 period crossover study design was conducted for 12 participants in Part 3)
Statistical Analysis 2: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — Treatment comparison (MK-8521 35μg - placebo) of the slope of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of the slope of ISR/G for MK-8521 35μg vs. placebo was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 2.67, 90% CI 2-sided [2.12 to 3.36]; [other analysis details as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg; Test type: Other — Treatment comparison (MK-8521 125μg - MK-8521 35μg) of the slope of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of the slope of ISR/G for MK-8521 125μg vs. MK-8521 35μg was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 1.73, 90% CI 2-sided [1.38 to 2.16]; [other analysis details as in outcome 31, analysis 1]

32. Secondary Outcome: Ratio of ISR/G at the Highest Glucose Infusion Rate During GGI Due to Treatment With A Single Dose of MK-8521 (Part 3)
Description: Pancreatic beta cell sensitivity to ambient glucose concentration after a single dose of MK-8521 125μg/35μg or placebo at Tmax was quantified as the ratio of the insulin secretion rate to glucose (ISR/G) at the highest glucose infusion rate during GGI (i.e., time weighted average between 120 to 160 minutes [TWA120-160min] of ratio [ISR/G]). Study drug was administered on Day -1 and blood concentrations of glucose, insulin, and C-peptide were determined at -10, -5 (pre-GGI), 20, 40, 60, 80, 100, 120, 140, and 160 minutes after start of GGI on Day 1 of each period.
Time Frame: From -10 to 160 minutes after GGI on Day 1
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: (ng/min)/(mg/dL)
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 11
(ng/min)/(mg/dL) | 0.0164 [0.0134 to 0.02] | 0.0256 [0.021 to 0.0312] | 0.0084 [0.0069 to 0.0103]
Statistical Analysis 1: Comparison: Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — Treatment comparison (MK-8521 125μg - placebo) of the ratio of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of TWA120-160min of ratio (ISR/G) for MK-8521 125μg vs. placebo was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 3.04, 90% CI 2-sided [2.62 to 3.53]; Number of participants included in analysis: N=17 (3-period crossover study design was conducted for 12 participants in Part 3)
Statistical Analysis 2: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 - Panel H - Placebo; Test type: Other — Treatment comparison (MK-8521 35μg - placebo) of the ratio of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of TWA120-160min of ratio (ISR/G) for MK-8521 35μg vs. placebo was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 1.94, 90% CI 2-sided [1.67 to 2.26]; [other analysis details as in outcome 32, analysis 1]
Statistical Analysis 3: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg; Test type: Other — Treatment comparison (MK-8521 125μg - 35μg) of the ratio of ISR/G during GGI at Tmax was performed using a linear mixed effect model with treatment and period as fixed effects and participant as random effect. The 90% confidence interval of GMR of TWA120-160min of ratio (ISR/G) for MK-8521 125μg - 35μg was calculated from the model; p < 0.001, Linear mixed effect model; Geometric mean ratio = 1.57, 90% CI 2-sided [1.35 to 1.82]; [other analysis details as in outcome 32, analysis 1]

33. Secondary Outcome: Glucose (TWA0-160min) During GGI at Tmax After a Single Dose of MK-8521 (Part 3)
Description: Glycemic effect during GGI after administration of a single dose of MK 8521 125mcg/35mcg or placebo at Tmax was evaluated as the time-weighted average of glucose concentration throughout the 160 minutes (TWA0-160min) of the GGI. Study drug was administered on Day -1 and blood glucose concentrations were determined at -10, -5 (pre GGI), 20, 40, 60, 80, 100, 120, 140, 160 minutes after start of GGI on Day 1 of each period. The parameter glucose (TWA0-160min) reflects ambient glucose concentration during the GGI.
Time Frame: From -10 to 160 minutes after GGI on Day 1
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 11
mg/dL | 118.38 [109.48 to 127.99] | 95.73 [88.84 to 103.16] | 147.94 [136.83 to 159.96]
Statistical Analysis 1: Comparison: Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 125mcg - placebo) in glucose (TWA0-160min) after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p < 0.001, Linear mixed effect model; Geometric mean ratio = 0.65, 90% CI 2-sided [0.6 to 0.7]; [other analysis details as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 - Panel H - Placebo; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 35μg - placebo) in glucose (TWA0-160min) after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p < 0.001, Linear mixed effect model; Geometric mean ratio = 0.8, 90% CI 2-sided [0.74 to 0.87]; [other analysis details as in outcome 32, analysis 1]
Statistical Analysis 3: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 125μg - MK-8521 35μg) in glucose (TWA0-160min) after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p < 0.001, Linear mixed effect model; Geometric mean ratio = 0.81, 90% CI 2-sided [0.75 to 0.87]; [other analysis details as in outcome 32, analysis 1]

34. Secondary Outcome: Maximum Glycemic Excursion (Gmax) During GGI and Tmax After a Single Dose of MK-8521 (Part 3)
Description: Glycemic effect during GGI after administration of a single dose of MK-8521 125μg/35μg or placebo at Tmax was evaluated as the Gmax during the GGI. Study drug was administered on Day -1 and blood glucose concentrations were determined at -10, -5 (pre-GGI), 20, 40, 60, 80, 100, 120, 140, and 160 minutes after start of GGI on Day 1 of each period. The parameter Gmax reflects ambient glucose concentration during the GGI.
Time Frame: From -10 to 160 minutes after GGI on Day 1
Population: as for outcome 21
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 11
mg/dL | 154.37 [136.5 to 174.48] | 120.43 [107.1 to 135.42] | 217.53 [192.35 to 246]
Statistical Analysis 1: Comparison: Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 125μg vs. placebo) in Gmax after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p < 0.001, Linear mixed effect model; Geometric mean ratio = 0.55, 90% CI 2-sided [0.49 to 0.63]; [other analysis details as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg vs Part 3 - Panel H - Placebo; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 35μg - placebo) in Gmax after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p < 0.001, Linear mixed effect model; Geometric mean ratio = 0.71, 90% CI 2-sided [0.62 to 0.81]; [other analysis details as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Part 3 Panel H MK-8521 35μg vs Part 3 Panel H MK-8521 125μg; Test type: Other — The least squares means and 90% confidence intervals for the treatment difference (MK-8521 125μg - MK-8521 35μg) in Gmax after a single dose was determined using a linear mixed effect model with treatment and period as fixed effects and participant as random effect; p = 0.004, Linear mixed effect model; Geometric mean ratio = 0.78, 90% CI 2-sided [0.69 to 0.89]; [other analysis details as in outcome 31, analysis 1]

35. Secondary Outcome: Area Under the Curve (AUC) 0-∞ for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 3)
Description: AUC0-∞ is a measure of the mean concentration levels of drug in the plasma after the dose. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part III [35 and 125 μg]) is presented. Method of dispersion is actually Coefficient of Variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. No pharmacokinetic data was available for AUC0-∞ for Part 3 due to sparse issues during the treatment period.
Time Frame: Day 1: predose, -60, -10 min pre-GGI, 40 min, 80 min, 120 min, 160 min, 360 min, and 600 min after start of GGI (Part 3)
Population: as for outcome 21
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: Area Under the Curve (AUC) 0-24hr. for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 3)
Description: AUC0-24hr is a measure of the mean concentration levels of drug in the plasma 0 to 24 hrs. after the dose. Mean pharmacokinetic parameter values for MK-8521 following administration of multiple subcutaneous once daily doses for 10 Days (with dose escalation on Day 5) to healthy non-obese male participants (Part II, Panel C, D, and E) are presented. Method of dispersion coefficient of variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. No pharmacokinetic data was available for AUC0-24hr. for Part 3 due to sampling issues during the treatment period.
Time Frame: as for outcome 35
Population: as for outcome 21
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Peak Plasma Concentration (Cmax) of Participants Treated With a Single Dose of MK-8521 (Part 3)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part III [35 and 125 μg]) is presented. Method of dispersion is actually Coefficient of Variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: as for outcome 35
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 0
nM | 0.418 (26.8) | 1.80 (21.7) |

38. Secondary Outcome: Time Taken to Reach Cmax (Tmax) for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 3)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the drug dose. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part III [35 and 125 μg]) is presented. No pharmacokinetic analysis was performed on participants receiving Placebo.
Time Frame: as for outcome 35
Population: as for outcome 21
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 11 | 12 | 0
Hours | 11.8 [11 to 18] | 12.7 [11 to 22] |

39. Secondary Outcome: Apparent Terminal Half-life (t1/2) for Plasma Concentration of Participants Treated With a Single Dose of MK-8521 (Part 3)
Description: Apparent Terminal Half-life (t1/2) is the time required for a given drug concentration in the plasma to decrease by 50%. A summary of pharmacokinetic parameters following administration of single SC (subcutaneous) injection of MK-8521 in healthy non-obese male participants (Part III [35 and 125 μg]) is presented. Method of dispersion is actually Coefficient of Variation (%CV). No pharmacokinetic analysis was performed on participants receiving Placebo. No pharmacokinetic data was available for t1/2 for Part 3 due to sampling issues during the treatment period.
Time Frame: Day 1: predose, -60, -10 min pre-GGI, 40 min, 80 min, 120 min, 160 min, 360 min, and 600 min after start of GGI(Part 3)
Population: as for outcome 21
Arm/Group | Part 3 Panel H MK-8521 35μg | Part 3 Panel H MK-8521 125μg | Part 3 - Panel H - Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The analysis population included all participants who received at least one dose of the investigational drug or placebo.
Groups:
- Part 1, Panel A, MK-8521 100μg: MK-8521 100μg in healthy male participants of 18 to 45 years of age
- Part 1, Panel A, MK-8521 300μg: MK-8521 300μg in healthy male participants of 18 to 45 years of age
- Part 1, Panel B, MK-8521 150μg: MK-8521 150μg in healthy male participants of 18 to 45 years of age
- Part 1, Panel B, MK-8521 175μg: MK-8521 175μg in healthy male participants of 18 to 45 years of age
- Part 1, Panel B, MK-8521 200μg: MK-8521 200μg in healthy male participants of 18 to 45 years of age
- Part 2, Panel C, MK-8521 50μg/72μg: MK-8521 50μg Days 1-5 and 72μg Days 6-10 or Placebo in healthy male participants of 18 to 45 years of age
- Part 2, Panel D, MK-8521 100μg/150μg: MK-8521 100μg Days 1-5 and 150μg Days 6-10 in healthy male participants of 18 to 45 years of age
- Part 2, Panel E, MK-8521 125μg/150μg: MK-8521 125μg Days 1-5 and 150μg Days 6-10 in healthy male participants of 18 to 45 years of age
- Part 2, Panel F, MK-8521 72μg/125μg: MK-8521 72μg Days 1-7 and 125μg Days 8-14 in obese male participants of 45 to 65 years of age
- Part 3, Panel H, MK-8521 35μg: MK-8521 35μg in healthy male participants of 18 to 45 years of age
- Part 3, Panel H, MK-8521 125μg: MK-8521 125μg in healthy male participants of 18 to 45 years of age
- Pooled Placebo: Placebo in healthy male participants of 18 to 45 years of age and obese male participants 45 to 65 years of age
Arm/Group | Part 1, Panel A, MK-8521 100μg | Part 1, Panel A, MK-8521 300μg | Part 1, Panel B, MK-8521 150μg | Part 1, Panel B, MK-8521 175μg | Part 1, Panel B, MK-8521 200μg | Part 2, Panel C, MK-8521 50μg/72μg | Part 2, Panel D, MK-8521 100μg/150μg | Part 2, Panel E, MK-8521 125μg/150μg | Part 2, Panel F, MK-8521 72μg/125μg | Part 3, Panel H, MK-8521 35μg | Part 3, Panel H, MK-8521 125μg | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/6 | 0/3 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/11 | 0/12 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/6 | 0/3 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/11 | 0/12 | 0/29
Other Adverse Events (participants affected / at risk) | 3/7 | 4/5 | 2/6 | 0/3 | 5/5 | 5/6 | 5/6 | 5/6 | 4/6 | 5/11 | 8/12 | 16/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1, Panel A, MK-8521 100μg (N=7) | Part 1, Panel A, MK-8521 300μg (N=5) | Part 1, Panel B, MK-8521 150μg (N=6) | Part 1, Panel B, MK-8521 175μg (N=3) | Part 1, Panel B, MK-8521 200μg (N=5) | Part 2, Panel C, MK-8521 50μg/72μg (N=6) | Part 2, Panel D, MK-8521 100μg/150μg (N=6) | Part 2, Panel E, MK-8521 125μg/150μg (N=6) | Part 2, Panel F, MK-8521 72μg/125μg (N=6) | Part 3, Panel H, MK-8521 35μg (N=11) | Part 3, Panel H, MK-8521 125μg (N=12) | Pooled Placebo (N=29)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 4 (4) | 2 (3) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.